CLINICAL TRIAL: NCT00358553
Title: A Crossover Study Assessing the Pharmacokinetics, Pharmacodynamics, and Safety of Recombinant Human Insulin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CT 101-002
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Last update posted 2007-03-13 (Estimated); Status verified 2007-03

CONDITIONS: Healthy
Keywords: Human Volunteers
MeSH Terms: interventions — Insulin

INTERVENTIONS:
Drug: Insulin

SUMMARY:
The purpose of this study is to assess the pharmacokinetics, pharmacodynamics, and safety of recombinant human insulin. The study will consist of 2 phases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male Subjects
* Age between 18 and 40 years of age

Exclusion Criteria:

* History of Diabetes
* Subjects with clinically significant active disease
* Known allergy to insulin

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, MD, Principal Investigator — Profil Institute
Locations (1):
- Profil, Neuss, Germany